CLINICAL TRIAL: NCT06298643
Title: Real-World Practice Patterns and Outcomes of Lower-Risk Myelodysplastic Syndrome Patients in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1094
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lower-risk Myelodysplastic Syndromes
MeSH Terms: interventions — Erythrocyte Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfusion dependent: Participants that received ≥2 units of red blood cell transfusion during the 8 weeks after initial myelodysplastic syndrome diagnosis date.
  Interventions: Procedure: Red blood cell transfusion
- Non-transfusion dependent: Participants that received 0 units or <2 units of red blood cell transfusion during the 8 weeks after initial myelodysplastic syndrome diagnosis date.
  Interventions: Procedure: Red blood cell transfusion

INTERVENTIONS:
Procedure: Red blood cell transfusion — ≥2 units of red blood cell transfusion
  Groups: Transfusion dependent
Procedure: Red blood cell transfusion — 0 units or <2 units of red blood cell transfusion
  Groups: Non-transfusion dependent

SUMMARY:
The purpose of this study is to describe the treatment patterns, clinical outcomes, healthcare resource utilization (HCRU) and medical costs of lower-risk myelodysplastic syndromes patients in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with at least one definitive myelodysplastic syndrome (MDS) diagnosis as per the 10th Revision of the International Statistical Classification of Diseases and Related Health Problems (MDS; ICD10: D46.X) between 01-May-2017 and 31-Jan-2022
* Participants with confirmed low-risk MDS by International Prognostic Scoring System (IPSS) or Revised International Prognostic Scoring System (IPSS-R) during baseline as follows:

  * Record of low (0 points) or intermediate-1 (>0 to 1 point) MDS according to IPSS scoring; or
  * Record of very low (≤1.5), low (>1.5-3), or intermediate (>3-4.5) MDS according to IPSS-R scoring; or
  * Mention of very low, low, intermediate, intermediate-1, or lower risk MDS in the Electronic Medical Records (EMR)
* Participants with a record of a confirmed bone marrow procedure (bone marrow aspiration code D404-00 and/or bone marrow biopsy code D404-02) during baseline period

Exclusion Criteria:

* Participants not meeting the inclusion criteria
* Participants <18 years of age at index date
* Participants who have a look back period <30 days from initial myelodysplastic syndrome diagnosis date

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult participants with myelodysplastic syndrome in Japan
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Participant age | At date of diagnosis
Participant sex | At date of diagnosis
Participant weight | At date of diagnosis
Participant height | At date of diagnosis
Participant comorbidities calculated using the Charlson Comorbidity Index (CCI) method | From 30 days prior to diagnosis up to 7 days post to diagnosis
Participant Eastern Cooperative Oncology Group (ECOG) score | From 30 days prior to diagnosis up to 7 days post to diagnosis
Participant International Prognostic Scoring System (IPSS) or Revised International Prognostic Scoring System (IPSS-R) risk category | Date of diagnosis, 6-months and 12 months post-diagnosis
Percentage of ring sideroblasts present in participants | Date of bone marrow test; from 30 days prior to diagnosis up to 7 days post to diagnosis
Percentage of bone marrow blasts present in participants | From 30 days prior to diagnosis up to 7 days post to diagnosis
Histopathology results | From 30 days prior to diagnosis up to 7 days post to diagnosis
Number of red-blood cell transfusions received by participants | Up to 56 days post diagnosis
Treatment prescribed by line of therapy | From date of diagnosis, up to 5-years
Duration of treatment by line of therapy | From date of diagnosis, up to 5-years
Time between date of diagnosis and treatment | From date of diagnosis to treatment initiation
Time between date of treatment initiation to treatment discontinuation | Date of treatment initiation, up to 5-years
Time between date of diagnosis to date of first red-blood cell transfusion | Date of diagnosis, up to 5-years

SECONDARY OUTCOMES:
Number of participants that achieved red-blood cell transfusion independence during first-line of therapy treatment | From week 1-24 and week 1-48 post date of treatment initiation
Mean hemoglobin change of participants during first-line of therapy | From week 1-24 and week 1-48 post date of treatment initiation
Number of transfusion dependant participants achieving re-blood cell transfusion independence for ≥12 weeks with associated concurrent mean hemoglobin increase of ≥1.5 g/dL during first-line of therapy | Week 1-24 post treatment initiation
Number of non-transfusion dependant participants achieving red-blood cell transfusion independence during first-line therapy for ≥24, 48 and 72 weeks | Week 24, 48 and 72 post date of initiation of treatment
Time to red-blood call transfusion independence of ≥12 weeks for transfusion dependant participants receiving first line therapy | From week 1-24 and week 1-48 post date of treatment initiation
Hematologic Improvement - Erythroid (HI-E) response of transfusion dependant participants receiving first line therapy | From week 1-24 post date of treatment initiation
Modified Hematologic Improvement - Erythroid (mHI-E) of transfusion dependant participants receiving first line therapy | From week 1-24 post date of treatment initiation
Hematologic Improvement - Erythroid (HI-E) response of non-transfusion dependant participants receiving first line therapy | From week 1-24 and week 1-48 post date of treatment initiation
Modified Hematologic Improvement - Erythroid (mHI-E) of non-transfusion dependant participants receiving first line therapy | From week 1-24 and week 1-48 post date of treatment initiation
Time to Hematologic Improvement - Erythroid (HI-E) or Modified hematologic improvement - Erythroid (mHI-E) during first-line therapy | From week 1-24 and week 1-48 post date of treatment initiation
Duration of Hematologic Improvement - Erythroid (HI-E) or Modified hematologic improvement - Erythroid (mHI-E) during first-line therapy | From date of treatment initiation to date of treatment discontinuation, up 5-years
Duration of red-blood call transfusion independence of ≥12 weeks for transfusion dependant participants receiving first line therapy | From date of treatment initiation to date of treatment discontinuation, up 5-years
Number of participants diagnosed with Acute Myeloid Leukemia | Date of treatment initiation, up to 5-years
Time to Acute Myeloid Leukemia diagnosis | Date of treatment initiation, up to 5-years
Overall survival (OS) of participants | 1, 2, 3 and 5-years post treatment initiation
Number of red-blood cell transfusion days per participant | Date of treatment initiation, up to 5-years
Number of red-blood cell units used per transfusion | Date of treatment initiation, up to 5-years
Number of outpatient visits per month | Date of treatment initiation, up to 5-years
Number of hospital admissions | Date of treatment initiation, up to 5-years
Length of hospitalization | Date of treatment initiation, up to 5-years
Reason for hospitalization | Date of treatment initiation, up to 5-years
Number of emergency department visits | Date of treatment initiation, up to 5-years
Number of Intensive care unit admissions (ICU) | Date of treatment initiation, up to 5-years
Number of outpatient/inpatient medication claims | Date of treatment initiation, up to 5-years
Supplemental medication use: Iron chelation use | Date of treatment initiation, up to 5-years
Supplemental medication use: Granulocyte-colony stimulating factors (G-CSF) | Date of treatment initiation, up to 5-years
Number of hematology tests ordered | Date of treatment initiation, up to 5-years
Medical costs | Date of treatment initiation, up to 5-years
  Including: cost of red-blood cell transfusion, cost of red-blood cell transfusion administration, cost of erythropoiesis stimulating agents (ESA) medication, cost of ESA administration, cost of iron chelation therapy medications, cost of iron chelation therapy administration, other costs and total costs

CONTACTS AND LOCATIONS:
Locations (1):
- Mebix, Inc, Tokyo, Minato-ku, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts